CLINICAL TRIAL: NCT00410072
Title: A Comparative Study of Chronic Hepatitis B Subjects Treated With Entecavir Plus Tenofovir Combination Therapy vs. Entecavir Monotherapy in Adults Who Are Treatment-Naive to Nucleosides and Nucleotides: The BE-LOW Study
Brief Title: Entecavir Plus Tenofovir Combination Therapy Versus Entecavir Monotherapy in Naive Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-110
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDF 0.5 mg (Experimental): TDF=tenofovir
  Interventions: Drug: Entecavir
- ETV 0.5 mg +TDF 300 mg (Experimental): ETV=entecavir; TDF=tenofovir
  Interventions: Drug: Entecavir + Tenofovir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, ETV = 0.5 mg, once daily, 100 weeks
  Other Names: Baraclude; BMS-200475
  Arms: TDF 0.5 mg
Drug: Entecavir + Tenofovir — Tablets, Oral, ETV = 0.5 mg + TFV = 300 mg, once daily, 100 weeks
  Other Names: Baraclude; BMS-200475
  Arms: ETV 0.5 mg +TDF 300 mg

SUMMARY:
The purpose of this study is to compare the effectiveness of entecavir plus tenofovir combination therapy with that of entecavir monotherapy. Safety will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B virus (HBV) infection (hepatitis B e antigen [HbeAg]-positive or negative) disease
* Nucleoside- and nucleotide-naive
* Males or females ≥16 years of age (or minimum age of consent in a given country)
* Compensated liver function
* HBV DNA >1.72*10*5*IU/mL (approximately 10*6*copies/mL) for HbeAg-positive participants
* HBV DNA >1.72*10*4*IU/mL (approximately 10*5*copies/mL) for Hbe-Ag-negative participants
* Alanine aminotransferase level ≥*upper limit of normal (ULN) and ≤10*ULN

Exclusion Criteria:

* Evidence of decompensated cirrhosis
* Coinfection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* Laboratory values out of protocol-specified range

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2007-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- United States (16):
  - Sergio E. Rojter, Los Angeles, California
  - Tuan Nguyen, Md, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - University Of Miami, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Digestive Healthcare Of Georgia, Atlanta, Georgia
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Maryland Digestive Disease Research, Llc, Laurel, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Sing Chan, Md, Flushing, New York
  - North Shore University, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Concorde Medical Group, New York, New York
  - Mount Sinai School Of Medicine, New York, New York
- Argentina (2):
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Rosario, Prov de Santa
- Australia (5):
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Prahan, Victoria
- Brazil (2):
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Porto Alegre Rs, Rio Grande do Sul
- Canada (4):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Toronto, Ontario
- France (4):
  - Local Institution, Grenoble
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Strasbourg
- India (4):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Lucknow
  - Local Institution, Ludhiana
  - Local Institution, Vellore
- Italy (4):
  - Local Institution, Antella Firenze
  - Local Institution, Brescia
  - Local Institution, Pisa
  - Local Institution, Roma
- Local Institution, Durango, Durango, Mexico
- Poland (5):
  - Local Institution, Bialystok
  - Local Institution, Chorzów
  - Local Institution, Krakow
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- South Africa (3):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Bellville, Western Cape
  - Local Institution, N1 City Goodwood, Western Cape
- Turkey (Türkiye) (4):
  - Local Institution, Bornova Izmir
  - Local Institution, Cebeci Ankara
  - Local Institution, Sihhiye Ankara
  - Local Institution, Trabzon

REFERENCES:
- [Derived] Lok AS, Trinh H, Carosi G, Akarca US, Gadano A, Habersetzer F, Sievert W, Wong D, Lovegren M, Cohen D, Llamoso C. Efficacy of entecavir with or without tenofovir disoproxil fumarate for nucleos(t)ide-naive patients with chronic hepatitis B. Gastroenterology. 2012 Sep;143(3):619-628.e1. doi: 10.1053/j.gastro.2012.05.037. Epub 2012 May 27. PMID 22643350
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 669 participants were enrolled; 384 were randomized. Among 285 who were not randomized, 266 did not meet the study criteria, 11 other, 1 poor compliance/noncompliance, 4 lost to follow-up, 1 withdrew consent, and 2 for administrative reasons.
Groups:
- ETV 0.5 mg: Entecavir (ETV) 0.5 mg monotherapy given once daily (QD) for 100 weeks
- ETV 0.5 mg +TDF 300 mg: ETV 0.5 mg plus Tenofovir (TDF) 300 mg combination therapy given QD for 100 weeks
Period: Day 1 to Week 48
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Started | 182 (Number of participants randomized and treated; 4 more were randomized but not treated.) | 197 (Number of participants randomized and treated; 1 more was randomized but not treated.)
Completed | 176 | 185
Not Completed | 6 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Other | 0 | 1
Not completed — poor compliance/noncompliance | 0 | 3
Not completed — Pregnancy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: After Week 48 to Week 96
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Started | 176 | 185
Completed | 170 | 174
Not Completed | 6 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Other | 2 | 0
Not completed — Poor compliance/noncompliance | 0 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg | Total
Number analyzed (Participants) | 182 | 197 | 379
Age, Customized [Number; unit: Participants]
  16 - 20 years | 13 | 19 | 32
  21 - 64 years | 157 | 169 | 326
  >=65 years | 12 | 9 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 51 | 117
  Male | 116 | 146 | 262
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 84 | 102 | 186
  Black/African American | 10 | 4 | 14
  Native Hawaiian/Other Pacific Islander | 1 | 1 | 2
  White | 83 | 87 | 170
  Other | 4 | 3 | 7
Country [Number; unit: participants]
  United States | 35 | 43 | 78
  Turkey | 11 | 11 | 22
  Russian Federation | 24 | 23 | 47
  Italy | 12 | 15 | 27
  India | 5 | 9 | 14
  France | 8 | 5 | 13
  Canada | 29 | 33 | 62
  Argentina | 12 | 15 | 27
  Poland | 15 | 13 | 28
  Brazil | 5 | 3 | 8
  Australia | 24 | 24 | 48
  South Africa | 2 | 3 | 5
Region [Number; unit: Participants]
  Africa | 2 | 3 | 5
  Asia | 29 | 33 | 62
  Europe | 70 | 67 | 137
  North America | 64 | 76 | 140
  South America | 17 | 18 | 35
Hepatitis B e antibody (HBeAb) at baseline [Number; unit: Participants]
  Positive | 60 | 60 | 120
  Negative | 122 | 137 | 259
Hepatitis B e antigen (HBeAg) status at baseline [Number; unit: Participants]
  Positive (> 172,000 IU/mL; approx 10^6 copies/mL) | 126 | 138 | 264
  Negative (> 17,200 IU/mL; approx 10^5 copies/mL) | 56 | 59 | 115
Hepatitis B surface antigen (HBsAg) status at baseline [Number; unit: Participants]
  Positive | 182 | 196 | 378
  Negative | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hepatitis B Virus DNA (HBV DNA) Levels <50 IU/mL by Polymerase Chain Reaction (PCR) at Week 96
Description: HBV DNA levels <50 IU/mL=approximately 300 copies/mL. Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Week 96
Population: Evaluable participants. A participant missing the efficacy assessments for a visit is considered a failure and is counted as evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants | 76.4 | 83.2
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Week 96; Test type: Superiority or Other; p = 0.0882, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [-1.0 to 14.9]

2. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Levels <50 IU/mL by PCR at Week 48 and Week 96 by Hepatitis B e Antigen (HBeAg) Status
Description: as for outcome 1
Time Frame: At Weeks 48 and 96
Population: Evaluable participants. If a participant is missing the efficacy assessments for a visit, this is considered a failure and is counted as evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants
  HBeAg+ at Week 48 (n=126, n=138) | 61.1 | 74.6
  HBeAg- at Week 48 (n=56, n=59) | 91.1 | 93.2
  HBeAg+ at Week 96 (n=126, n=138) | 69.8 | 80.4
  HBeAg- at Week 96 (n=56, n=59) | 91.1 | 89.8
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 13.5, 95% CI 2-sided [2.3 to 24.8]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-7.7 to 12.0]
Statistical Analysis 3: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Test type: Superiority or Other; p = 0.0460, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.6, 95% CI 2-sided [0.2 to 21.0]
Statistical Analysis 4: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-12.0 to 9.5]

3. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Levels <LOQ by PCR at Weeks 48 and 96
Description: LOQ=lower limit of quantitation. LOQ=29 IU/mL, or approximately 169 copies/mL. LOQ is the level above which quantitative results may be obtained with a specified degree of confidence. The LOQ is mathematically defined as equal to 10 times the standard deviation of the results for a series of replicates used to determine a justifiable limit of detection. Limits of quantitation are matrix-, method-, and analyte-specific.Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Weeks 48 and 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants
  Overall at Week 48 | 67.6 | 74.6
  Overall at Week 96 | 74.7 | 81.7
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at week 48. The stratified analysis was based on HBeAg strata at randomization; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [-1.8 to 16.0]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at week 96. The stratified analysis was based on HBeAg strata at randomization; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [-1.1 to 15.2]

4. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Levels <LOD by PCR at Weeks 48 and 96
Description: LOD=Lower limit of detection. LOD) LOD=10 IU/mL, or approximately 58 copies/mL. LOD is the lowest concentration level that can be determined to be statistically different from a blank (99% confidence). The LOD is typically determined to be in the region where the signal to noise ratio is greater than 5. Limits of detection are matrix-, method-, and analyte-specific.Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Weeks 48 and 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants
  Overall at Week 48 | 58.2 | 66.0
  Overall at Week 96 | 68.1 | 76.6
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48. The stratified analysis was based on HBeAg strata at randomization; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-1.5 to 17.1]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96. The stratified analysis was based on HBeAg strata at randomization; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [-0.2 to 17.3]

5. Secondary Outcome: Mean Log 10 HBV DNA at Weeks 48 and 96
Description: HBV DNA was analyzed by PCR, using the Roche COBAS®TaqMan - HPS assay. Reduction in Log 10 HBV count=reduced viral load.
Time Frame: Baseline, Weeks 48 and 96
Population: Evaluable participants at given time point. If a participant is missing the efficacy assessments for a visit, this is considered a failure and is counted as evaluable.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
log10 copies/mL
  Baseline (n=182, 197) | 7.48 (0.109) | 7.53 (0.100)
  Overall at Week 48 (n=176, 180) | 1.88 (0.065) | 1.56 (0.026)
  Overall at Week 96 (n=165, 170) | 1.68 (0.048) | 1.51 (0.038)

6. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Weeks 48 and 96
Description: ALT normalization= ≤1*upper limit of normal (ULN). Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Weeks 48 and 96
Population: Evaluable participants. A participant missing the efficacy assessments for a visit is considered a failure and counted as evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants
  Overall at Week 48 | 83.0 | 72.6
  Overall at Week 96 | 81.9 | 68.0
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48. The stratified analysis is based on HBeAg strata at randomization; Test type: Superiority or Other; NC+F; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-18.8 to -2.0]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96. The stratified analysis is based on HBeAg strata at randomization; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-21.5 to -4.1]

7. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss at Weeks 48 and 96
Description: HBeAg is a hepatitis B viral protein and is an indicator of active viral replication. Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Weeks 48 and 96
Population: Treated HBeAg-positive participants. If a participant was missing the efficacy assessments for a visit, this is considered a failure and was counted as evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 126 | 138
Percentage of participants
  Week 48 | 25.4 | 19.6
  Week 96 | 3.97 | 29.7
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-15.9 to 4.2]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -9.2, 95% CI 2-sided [-20.6 to 2.3]

8. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion [( at Weeks 48 and 96
Description: HBeAg seroconversion=HBeAg loss and presence of hepatitis B e antibody (HBeAb). HBeAg is a hepatitis B viral protein and is an indicator of active viral replication.
Time Frame: At Weeks 48 and 96
Population: Treated HBeAg-positive participants. A participant missing the efficacy assessments for a visit was considered a failure and was counted as evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 126 | 138
Percentage of participants
  Week 48 | 22.2 | 18.1
  Week 96 | 32.5 | 21.7
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-13.8 to 5.6]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-21.5 to -0.1]

9. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Weeks 48 and 96
Description: HBsAg = A part of the hepatitis B virus. When found in the blood, HBsAg is an early marker of infection. Analyses of binary efficacy endpoint during on-treatment period focused on participants who received treatment and used the analysis of noncompleter=failure (NC=F). All participants who received treatment were included in the denominator, and participants with missing measurements were counted as nonresponders for the specific endpoints.
Time Frame: At Weeks 48 and 96
Population: as for outcome 7
Measure: Number; unit: Percent of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 126 | 138
Percent of participants
  Week 48 | 3.2 | 1.4
  Week 96 | 4.0 | 5.1
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-5.3 to 1.9]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-3.9 to 6.1]

10. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Weeks 48 and 96
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection.
Time Frame: At Weeks 48 and 96
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 126 | 138
Percentage of participants
  Week 48 | 0.8 | 0.7
  Week 96 | 1.6 | 2.9
Statistical Analysis 1: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 48; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.2 to 2.0]
Statistical Analysis 2: Comparison: ETV 0.5 mg vs ETV 0.5 mg +TDF 300 mg; Analysis at Week 96; Test type: Superiority or Other; NC=F; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.3 to 4.9]

11. Secondary Outcome: Number of Participants With HBV DNA in Relevant Categories at Weeks 48 and 96
Description: Using the Roche COBAS TaqMan - HPS assay. Lower limit of Quantitation (LOQ) is the level above which quantitative results may be obtained with a specified degree of confidence. The LOQ is mathematically defined as equal to 10 times the standard deviation of the results for a series of replicates used to determine a justifiable limit of detection. Limits of quantitation are matrix-, method-, and analyte-specific.
Time Frame: At Weeks 48 and 96
Population: All treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Percentage of participants
  < LOQ (29 IU/mL) at Week 48 | 67.6 | 74.6
  LOQ - <50 IU/mL at Week 48 | 2.7 | 5.6
  50 - <172 IU/mL at Week 48 | 7.1 | 6.6
  172 - <1720 IU/mL at Week 48 | 7.7 | 4.1
  1720 - <17,200 IU/mL at Week 48 | 9.3 | 0.5
  17,200 - <172,000 IU/mL at Week 48 | 1.6 | 0
  ≥172,000 IU/mL at Week 48 | 0.5 | 0
  Missing at Week 48 | 3.3 | 8.6
  < LOQ (29 IU/mL) at Week 96 | 74.7 | 81.7
  LOQ - <50 IU/mL at Week 96 | 1.6 | 1.5
  50 - <172 IU/mL at Week 96 | 3.3 | 1.0
  172 - <1720 IU/mL at Week 96 | 5.5 | 1.5
  1720 - <17,200 IU/mL at Week 96 | 4.9 | 0
  17,200 - <172,000 IU/mL at Week 96 | 0.5 | 0
  ≥172,000 IU/mL at Week 96 | 0 | 0.5
  Missing at Week 96 | 9.3 | 13.7

12. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, and Discontinuations From Study Drug Due to Adverse Events or Laboratory Abnormalities
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded.
Time Frame: From enrollment through Week 100 + 24-week follow-up
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 182 | 197
Participants
  Deaths | 0 | 3
  SAEs | 12 | 14
  Adverse events | 132 | 131
  Discontinuations due to AEs | 2 | 5
  Related AEs | 39 | 49

13. Secondary Outcome: Number of Participants With HBV Resistance Through Week 48
Description: ETVr=entecavir resistance; TDFr=tenofovir resistance. HBV polymerase using the Trugene® HBV Genotyping Kit. HBV resistance: genotyping of HBV polymerase will be performed on stored viral samples at any timepoint when considered appropriate based on virologic response, including any specimen with detectable HBV DNA. When appropriate, phenotyping will also be used.
Time Frame: Week 48
Population: All participants who received study drug and with HBV DNA levels >=50 IU/mL
Measure: Number; unit: Participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 51 | 33
Participants
  ETVr | 0 | 0
  TDFr | 0 | 0

14. Secondary Outcome: Number of Participants With HBV Resistance at Week 96
Description: ETVr=entecavir resistance; TFDr=tenofovir resistance. HBV polymerase using the Trugene® HBV Genotyping Kit. HBV resistance: genotyping of HBV polymerase will be performed on stored viral samples at any timepoint when considered appropriate based on virologic response, including any specimen with detectable HBV DNA. When appropriate, phenotyping will also be used.
Time Frame: Week 96
Population: Participants who received study drug and with HBV DNA levels >=50 IU/mL.
Measure: Number; unit: Participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 33 | 10
Participants
  ETVr | 0 | 0
  TDFr | 0 | 0

15. Secondary Outcome: Number of Participants With Virologic Breakthrough at Week 48
Description: ETVr=entecavir resistance; TFDr=tenofovir resistance. Virologic breakthrough= confirmed >= 1 log10 increase in HBV DNA from the on-treatment nadir
Time Frame: Week 48
Population: Participants with confirmed >=1 log10 increase in HBV DNA from the on-treatment nadir
Measure: Number; unit: Participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 1 | 7
Participants
  ETVr | 0 | 0
  TDFr | 0 | 0

16. Secondary Outcome: Number of Participants With Virologic Breakthrough at Week 96
Description: ETVr=entecavir resistance; TFDr=tenofovir resistance. Virologic breakthrough=confirmed >=1 log10 increase in HBV DNA from moving nadir
Time Frame: Week 96
Population: Participants with confirmed >= 1 log10 increase in HBV DNA from moving nadir
Measure: Number; unit: Participants
Arm/Group | ETV 0.5 mg | ETV 0.5 mg +TDF 300 mg
Number analyzed (Participants) | 1 | 7
Participants
  ETVr | 0 | 0
  TDFr | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to Week 100 (on study), Post-dosing follow-up - 24 Weeks
Description: Participants who have study medication completed or discontinued permanently were followed for 24 weeks post-dosing for safety.
Groups:
- ETV 0.5 mg: ETV 0.5 mg monotherapy given QD for 100 weeks
- ETV/TDF 0.5 mg +TDF 300 mg: ETV 0.5 mg plus TDF 300 mg combination therapy given once daily (QD) for 100 weeks
Arm/Group | ETV 0.5 mg | ETV/TDF 0.5 mg +TDF 300 mg
Serious Adverse Events (participants affected / at risk) | 13/182 | 14/197
Other Adverse Events (participants affected / at risk) | 69/182 | 73/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETV 0.5 mg (N=182) | ETV/TDF 0.5 mg +TDF 300 mg (N=197)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1
HEPATITIS (Hepatobiliary disorders) | 0 | 1
HEPATITIS A (Infections and infestations) | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEPATITIS B (Infections and infestations) | 0 | 1
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 1
BLOOD AMYLASE INCREASED (Investigations) | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETV 0.5 mg (N=182) | ETV/TDF 0.5 mg +TDF 300 mg (N=197)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 | 9
DIARRHOEA (Gastrointestinal disorders) | 11 | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 13
FATIGUE (General disorders) | 11 | 12
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 8
HEADACHE (Nervous system disorders) | 19 | 22
NAUSEA (Gastrointestinal disorders) | 9 | 20
NASOPHARYNGITIS (Infections and infestations) | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication